CLINICAL TRIAL: NCT07254338
Title: Blood and uRine Metabolomics Exploration for Assessing Thoracic Health After Treatment of Group 3 Pulmonary Hypertension
Brief Title: Exploration of Metabolome in Patients With Interstitial Lung Disease and Pulmonary Hypertension With or Without Specific Pulmonary Hypertension Treatment
Acronym: BREATH-TPT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0216
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Lung Disease; Precapillar Pulmonary Hypertension
Keywords: ILD-PH; Inhaled Treprostinil; PH treatment; Metabolomic
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (veinous) collected under standard care conditions, in a dry red blood tube without additional gel (4 mL) to obtain serum after centrifugation for 10 minutes at 1500g, in the form of 500µL aliquots. Blood samples will be collected at inclusion and at completion.
  Urine collected from patient into a dry powder compact in the waiting room before or after the consultation. Preparation of two cryotubes containing at least 1 mL per sample, labelled with the patient's code in the study. Hospital urine samples will be taken at inclusion, once during early follow-up, and a final time at the end of follow-up.
  Furnitures will be given to patients to match clinical condition for auto-sampling for those who will accept to make the samples at home. 1 auto-sample every two weeks, 6 times between inclusion and the end of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group "intervention": Patients who suffer from ILD and ILD-PH from this group will be given specific treatments (especially inhaled TREPROSTINIL, up to 3 breath per use; 4 uses a day) for ILD-PH after usual independent collegial consultation Those patients will have before and after treatment blood and urine metabolomic profile.
  They will have baseline and follow up blood and urine sampling. They will be offer possibility to perform up to 6 auto-sampling at home.
  Interventions: Other: Blood sampling for metabolomic profiling; Other: Urine sampling for metabolomic profiling
- Group " control ": Patients who suffer from ILD and ILD-PH from this group will not be given specific ILD-PH treatment based on insufficient haemodynamic data or clinical contraindications after independent collegial consultation.
  They will have only baseline blood and urine sampling.
  Interventions: Other: Blood sampling for metabolomic profiling; Other: Urine sampling for metabolomic profiling

INTERVENTIONS:
Other: Blood sampling for metabolomic profiling — Blood (veinous) will be collected under standard care conditions, in a dry red blood tube without additional gel (4 mL) to obtain serum after centrifugation for 10 minutes at 1500g, in the form of 500µL aliquots, labelled with the patient's code in the study.
  This sampling will be performed at baseline in both group; and after follow up completion in Group 1 (4-6 month)
Other: Urine sampling for metabolomic profiling — Urine collected from patient into a dry powder compact in the waiting room before or after the consultation. Preparation of two cryotubes containing at least 1 mL per sample, labelled with the patient's code in the study. In the absence of a calling point, strict aseptic conditions are not required, as the use of chemicals or antiseptic soaps can interfere with the dosages.
  This sampling will be performed in Group 1 and 2 at baseline; and in Group 1 at 2-month and after completion of follow-up time (4-6 month).

SUMMARY:
Fibrosing interstitial lung diseases (FILDs) encompass a group of rare diseases characterized by progressive pulmonary fibrosis leading to respiratory failure. Current treatments primarily aim to slow disease progression but remain limited, making lung transplantation the ultimate recourse.

The development of pulmonary hypertension (PH) in the context of FILDs significantly worsens morbidity and mortality and drastically reduces patients' life expectancy. Conventional treatments for PH are generally ineffective in this setting. Nevertheless, some promising therapeutic agents are currently under investigation, particularly inhaled prostacyclin analogs such as treprostinil, which have demonstrated efficacy in recent clinical studies.

Our study aims to explore, in a minimally invasive manner, variations in metabolites in the serum and urine of patients with PH secondary to FILDs, before and during treatment. The main objective is to better understand the systemic effect of these treatments. Furthermore, the identification of metabolomic signatures will allow us to differentiate responders from non-responders, thus providing valuable prognostic and predictive criteria.

To date, some patients do not benefit from the available treatments, and better selection of responders could prevent iatrogenic effects in patients whose clinical condition is already fragile. In addition, characterizing the systemic mode of action of these treatments could pave the way for new clinical research focused on the profiles of responding patients.

Finally, a thorough understanding of the efficacy of the studied therapies is essential. Indeed, effective treatment of PH in the context of FILDs could not only slow disease progression but also reduce the need for lung transplantation, a major challenge in a context of organ shortage.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from progressive interstitial lung disease (ILD) and especially lung fibrosis
* Suspicion of precapillar pulmonary hypertension (group 3 PH / ILD-PH)
* Patients undergoing cardiac catheterisation for haemodynamic confirmation
* Patient who has given informed consent

Exclusion Criteria:

* Patients suffering from other forms of PH (i.e. PAH, CTEPH, heart failure, multifactorial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients monitored at Hospices Civils de Lyon for Interstitial Lung Disease, with suspected group 3 PH, for whom the medical team is considering or discussing the indication for specific ILD-PH treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of urinary metabolite concentrations before and after initiation of treatment measured centrally by proton nuclear magnetic resonance spectroscopy (¹H-NMR). | Outcome is measured when all patients will have their 4-6 months follow-up completed.
  The 1H-NMR analysis of each patient's urine will enable us to obtain a table showing the absolute concentration of metabolites per individual.
  The effects of the drug response will be interpreted following pairwise-comparisons of metabolite concentrations per individual within Group 1, and expressed as fold change to perform a pathway assessment, notably using Metabo Analyst tool
Comparison of blood metabolite concentrations before and after initiation of treatment measured centrally by proton nuclear magnetic resonance spectroscopy (¹H-NMR). | Outcome is measured when all patients will have their 4-6 months follow-up completed.
  The 1H-NMR analysis of each patient's blood will enable us to obtain a table showing the absolute concentration of metabolites per individual.
  The effects of the drug response will be interpreted following pairwise-comparisons of metabolite concentrations per individual within Group 1, and expressed as fold change to perform a pathway assessment, notably using Metabo Analyst tool.
  It will also allow us to explore kidney filtration effect on metabolic profile
Comparative prognosis analysis within sub-groups | Outcome is measured when all patients will have their 4-6 months follow-up completed.
  Based on clinical response, several subgroups will be defined (responders, non-responders, paradoxical worsening) in order to define prognostic signatures using intergroup statistical comparisons of baseline metabolic concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cardiologique et Pneumologique Louis Pradel, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No